CLINICAL TRIAL: NCT00539851
Title: Risk Factors for Developing Diabetes Mellitus After Allogenic Stem Cell Transplantation
Brief Title: Risk Factors for Diabetes After Stem Cell Transplantation
Status: Completed | Type: Observational
Sponsor: Vanderbilt University (Other)
Collaborators: Sanofi (Industry)
Responsible Party: Shubhada Jagasia, MD, Vanderbilt University Medical Center
Other Study IDs: #040639
Record Dates: First submitted 2007-10-04; First posted 2007-10-05 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2010-03

CONDITIONS: Diabetes Mellitus
Keywords: Allogenic Stem Cell Transplantation; Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is proposed to investigate the incidence of Post Transplant Diabetes Mellitus (PTDM) as well as associated risk factors for the development of PTDM in patients undergoing allogenic stem cell transplantation.

DETAILED DESCRIPTION:
Allogenic stem cell transplantation from related or unrelated donors has been used successfully to cure patients with a variety of hematological malignancies. Graft-versus-host disease (GVHD) is an alloreactive immune phenomenon, where the activated donor T cells recognizes the recipient as being foreign and effects a cytotoxic response. GVHD occurring in the first 100 days after transplantation is termed acute GVHD and is characterized by hepatitis, dermatitis, and enteritis.

High dose corticosteroids remain one of the cornerstone therapies to treat acute GVHD. However, an association between corticosteroid therapy and the development of diabetes mellitus after solid organ transplantation has become widely recognized. Similarly, post transplant diabetes mellitus (PTDM) has been increasingly noted in the allogenic stem cell transplant population, however, to date, no systematic study has been completed to identify the incidence of PTDM and associated risk factors. We propose to investigate the incidence of PTDM as well as associated risk factors for the development of PTDM in patients undergoing allogenic stem cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 65 years or age
* Fulfills institutional criteria for and is scheduled to undergo an allogenic stem cell transplantation at VUMC

Exclusion Criteria:

* Younger than 18 years or older than 65 years
* Pre-existing diabetes mellitus
* Positive pregnancy test
* Unable to complete the conditioning regimen prior to stem cell transplantation
* Unable to give informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients will be enrolled through the Endocrinology, Hematology and Stem Cell Transplantation Clinics at Vanderbilt University Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2005-11; Primary Completion 2009-08 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shubhada Jagasia, MD, Principal Investigator — Vanderbilt University Medical Center